CLINICAL TRIAL: NCT05302024
Title: Efficacy and Safety of Iguratimod in the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia: a Phase 2, Open-label, Single-arm Trial
Brief Title: Efficacy and Safety of Iguratimod in the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-ITP 001
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — iguratimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iguratimod treatment (Experimental): Iguratimod is given at a dose of 25 mg bid for 12 weeks.
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — Oral iguratimod (25 mg twice daily) for 12 weeks. Iguratimod is a new drug for the treatment of rheumatoid arthritis (RA) and osteoarthritis (OA), which was filed for marketing in Japan in 2003. It can significantly reduce the inflammatory response, not only selectively inhibit COX-2, but also inhibit the production of inflammatory cytokines, tumor necrosis factor, lymphocytes and immunoglobulins, and has an autoimmunomodulatory effect; it has a rapid onset of action, better efficacy and fewer adverse effects than existing drugs, and is effective in patients for whom other drugs are ineffective. It has been reported in the literature that in vitro iguratimod can inhibit the activity of nuclear factor-κB (NF-κB), which in turn inhibits the production of inflammatory cytokines (interleukin-1, interleukin-6, interleukin-8, tumor necrosis factor alpha). Iguratimod also interacts directly with mouse and human B cells in vitro to inhibit the production of immunoglobulins.

SUMMARY:
A phase 2, open-label, single-arm study to evaluate the efficacy and safety of iguratimod for the treatment of adults with steroid-resistant/relapse immune thrombocytopenia (ITP)

DETAILED DESCRIPTION:
The investigators are undertaking an open-label, single-arm study of 100 adults with steroid-resistant/ relapse ITP in China. Patients were received Iguratimod treatment. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* 18 years older;

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* Congestive heart failure
* Severe arrhythmia
* Nursing or pregnant women
* Aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
* Creatinine or serum bilirubin levels each 1•5 times or more than the normal range
* Active or previous malignancy
* Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-22 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Durable response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Initial response | 1 month
  Platelet count ≥ 30 x 10^9/L and at least doubling baseline at 1 month
Remission | 12 months
  109/ Platelet count >100x 10^9/L at 12 mon
Time to response | 12 months
  Time to response was defined as the time from starting treatment to the time to achieve the response
Bleeding | 12 months
  Major bleeding: (1) WHO grade 3 or 4 bleeding, (2) Buchanan severe grade, (3) Bolton-Maggs and Moon "major bleeding," (4) IBLS grade 2 or higher, or (5) life-threatening or intracerebral hemorrhage bleeding
Adverse events | 12 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No